CLINICAL TRIAL: NCT05852158
Title: The Use of Single Dose vs Short-Term Peri-Operative Cefazolin in the Prevention of Surgical Site Infection Following Orthognathic Surgery
Brief Title: Antibiotics for Prevention of Infection Following Orthognathic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Abdul El-Rabbany (Other)
Responsible Party: Sponsor-Investigator, Abdul El-Rabbany, Principal Investigator, Oral and Maxillofacial Surgery Resident, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1028749
Record Dates: First submitted 2023-04-10; First posted 2023-05-10 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Orthognathic Surgical Site Infection
Keywords: Orthognathic Surgery; Surgical Site Infection; Peri-Operative Antibiotics; Post-Operative Antibiotics; Pre-Operative Antibiotics; Antibiotic Prophylaxis; Cefazolin
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefazolin

STUDY DESIGN:
Intervention Model Description: Our plan is to conduct a prospective, randomized controlled trial evaluating patients undergoing orthognathic surgery including bilateral sagittal split osteotomies with or without concomitant maxillary and/or chin surgery, with or without wisdom teeth extraction. All patients meeting the inclusion criteria will be offered participation, and informed consent will be obtained at the pre-operative appointment following surgical consent. The patients will then be assigned a study number and randomly allocated to one of two groups as follows:
  A) Single pre-operative dose of 2g IV Cefazolin B) Single pre-operative dose of 2g IV Cefazolin followed by a 24-hour course of 2g IV Cefazolin every 8 hours All patients will receive the same post-operative instructions and will be discharged with 0.12% chlorhexidine mouth rinse to be used for 2 weeks following discharge. Patients will return for follow-up at 2 weeks, 4 weeks, and 6 weeks following discharge.
Who Masked: Outcomes Assessor
Masking Description: Surgeons assessing for the presence of surgical site infection will be blinded to the antibiotic regimen that the patient received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single Dose (Experimental): Single pre-operative dose of 2g IV Cefazolin given prior to first incision for orthognathic surgical procedure
  Interventions: Drug: Cefazolin 2 GM Injection
- 24-Hour Dosing (Active Comparator): Single pre-operative dose of 2g IV Cefazolin given prior to first incision for orthognathic surgical procedure, as well as 2g IV Cefazolin q8h post-operatively for 24 hours (3 total doses)
  Interventions: Drug: Cefazolin Injection

INTERVENTIONS:
Drug: Cefazolin 2 GM Injection — Single pre-op dose of 2g IV cefazolin
  Other Names: Single Dose IV Cefazolin
  Arms: Single Dose
Drug: Cefazolin Injection — Pre-op dose of 2g IV cefazolin along with 3 post-op doses of 2g IV cefazolin every 8 hours
  Other Names: Four Doses IV Cefazolin
  Arms: 24-Hour Dosing

SUMMARY:
Orthognathic surgery describes a group of procedures aimed at correcting developmental or acquired deformities of the jaws and facial skeleton. The goal of these procedures is to improve speech, jaw and dental function, aesthetics, and symptoms of sleep apnea. This is accomplished by surgical repositioning of the upper jaw (maxilla) and lower jaw (mandible). The most common procedures are lefort I osteotomies (upper jaw repositioning) and bilateral sagittal split osteotomies (lower jaw repositioning). At our institution, almost all cases include one or both of these two procedures. The majority of cases include bilateral sagittal split osteotomies (BSSO). As access to the jaws is through the oral cavity, these procedures are considered to be clean-contaminated surgeries due to the high intra-oral bacterial load. The result is that surgical site infections (SSIs) occur in 10-15% of cases. Studies show that the vast majority of these infections occur in the lower jaw (BSSO sites), presumably due to pooling of saliva and debris. SSIs are associated with patient discomfort, prolonged hospital stays, increased morbidity, and increased cost to healthcare systems.

The use of peri-operative antibiotics has been shown to significantly reduce the incidence of SSI following orthognathic surgery. There is currently no consensus on the dosing or specific antibiotic to be used. There is strong evidence that pre-operative antibiotics significantly decrease SSI compared to no antibiotics. However, to date, there is no good evidence to support the use of post-operative antibiotics to further decrease the rate of infection. Several studies have examined the use of post-operative antibiotics ranging between 1-7 days. The majority of studies were not able to demonstrate a statistically significant difference to justify the use of post-operative antibiotics. A systematic review by Danda and Ravi in 2011 suggested that there likely is a benefit to the use of post-operative antibiotics. Danda and colleagues in 2017 later conducted a trial comparing pre-operative antibiotics alone compared to pre-operative combined with post-operative antibiotics. A statistically significant difference was not found, however, they felt that this was due to a limited sample size. Overall, there is no robust data that supports the use of post-operative antibiotics. The World Health Organization guidelines currently recommend against the use of post-operative antibiotics in orthognathic surgery. However, they do comment that there is some weak evidence that suggests its use. It was deemed that this low quality evidence did not outweigh the potential harm of antimicrobial resistance, which results from inappropriate overuse of antibiotics. Antimicrobial resistance is a serious, growing problem which has deadly consequences.

Our current protocol at the QEII Health Sciences Center for peri-operative antibiotic administration is a single pre-operative dose of 2g cefazolin IV, followed by further doses every 8 hours post-operatively for a total of 24 hours (3 post-operative doses). Our study aims to investigate whether there is a need for these additional post-operative doses. If there is a benefit to these additional doses, the research team aims to investigate whether this benefit outweighs the risks. This question is of great importance in order to avoid an unnecessary contribution to antibiotic resistance and unnecessary potential adverse effects.

Participants will be assigned a study number and randomly allocated to one of two groups. Group A will receive a single pre-operative dose of 2g IV cefazolin. Group B will receive a pre-operative dose of 2g IV cefazolin, followed by an additional three doses post-operatively every 8 hours for a total of 24 hours.

Informed consent will be obtained at each participant's pre-operative assessment in the days leading up to the procedure. The participant will then select a group designation from a sufficiently mixed jar, and group A or B will be assigned to their study number.

For each patient, the procedures completed will be documented, along with age, sex, smoking status, length of procedures, and complications. Complications including medication adverse reaction (allergy, toxicity, side effects), surgical complications, and any other significant complications related to the medications or deemed to be relevant to infection risk will be documented. Procedures will be carried out in the standard fashion. Patients will receive the same post-operative instructions and will be discharged with a chlorhexidine mouth rinse to be used for two weeks. Patients will return for follow-up at 2 weeks, 4 weeks, and 6 weeks post-operatively. Surgical site infection diagnosis will be made according to the CDC criteria and will be reported as either superficial, deep, or organ/space infections. Date of occurrence, location of infection, and treatment provided will be recorded on a standard form provided to surgeons.

DETAILED DESCRIPTION:
Background

Orthognathic surgery describes a group of procedures whose main goal is to correct congenital and acquired dentofacial deformities, thereby improving speech, mastication, aesthetics, and symptoms of sleep apnea. These outcomes may be achieved by surgical repositioning of the maxilla and mandible using a variety of methods, the most common being Lefort I osteotomies, bilateral sagittal split osteotomies, intraoral vertical ramus osteotomies, and functional genioplasty. As access for these methods involves trans-oral approaches, these procedures are considered to be clean-contaminated surgeries due to the high intra-oral bacterial load. As a result, surgical site infection (SSI) rates are reported in the literature to range from 10-15% following orthognathic surgery. SSIs are associated with patient discomfort, prolonged hospital stays, increased morbidity, and increased cost to healthcare systems.

The use of peri-operative antibiotics has been demonstrated to significantly reduce the incidence of SSI following orthognathic surgery. However, there is continued debate regarding the most effective antibiotic protocol, and no consensus regarding timing or specific antibiotic has been achieved. A 1999 study conducted demonstrated a significant difference in SSI rates between patients treated with a single pre-operative dose of antibiotics compared to placebo. A systematic review in 2011 reported that there likely is a benefit to the use of post-operative antibiotics extended for 1-7 days versus a single pre-operative dose. Antibiotic course length was further evaluated in 2016, the investigators demonstrated a significant difference in effectiveness of 3-day courses of antibiotics vs 1-day. However, the number needed to treat was 10, due to which the conclusion was made that the potential harms may not outweigh the risks. Several studies conducted have failed to justify the prolonged use of post-operative antibiotics past 24 hours. As such, it seems that the common standard is the use of pre-operative antibiotics in conjunction with short-term (24-hours or less) post-operative antibiotic courses. To date, few studies have been conducted comparing SSI rates in patients receiving a single pre-operative antibiotic dose to those in patients receiving a pre-operative dose in conjunction with a 24-hour post-operative course. A trial conducted in 2017 found an SSI rate of 9.3% in patients receiving a single pre-operative antibiotic dose compared to 2.6% in patients receiving a pre-operative dose in conjunction with a 24-hour post-operative course, however, the results were not statistically significant. The group attributed this result to an inadequate sample size. In a 2013 study, researchers demonstrated a significant difference in SSI rate between patients receiving a single dose of pre-operative intravenous (IV) Amoxicillin compared to those receiving an additional two doses post-operatively. This, however, is in contrast to several studies which failed to demonstrate a benefit of post-operative antibiotics compared to single pre-operative doses. Overall, there seems to be no robust data supporting the use of post-operative antibiotics following orthognathic surgery. With limited data supporting prolonged antibiotic use, one must question if there are any benefits to offset the risks of antibiotic over-use, which include medication adverse effects, increased healthcare costs, and most importantly, antibiotic resistance. The World Health Organization (WHO) published guidelines recommend no prolongation of antibiotic administration post-operatively following orthognathic surgery, as it was deemed that the low quality evidence supporting its use did not outweigh the potential harm of antimicrobial resistance.

In addition to course length and timing, the choice of antibiotic also plays a major role in SSI rate following orthognathic surgery. The most commonly reported antibiotics used in clinical trials appear to be penicillin, amoxicillin, cefazolin, clindamycin, and ampicillin. A systematic review was conducted in 2019, which reported improved efficacy of cefazolin compared to clindamycin and penicillin in preventing post-orthognathic surgery SSIs.

The most common bacterial isolates from odontogenic infections are Viridans group streptococci, Peptostreptococcus, Prevotella, Fusobacterium, and Bacteroides. Overall, cefazolin has high susceptibility rates against the most common oral bacteria. Cefazolin shows excellent susceptibility rates against Viridans group streptococci, Peptostresptococcus, Prevotella, and Fusobacterium.

The purpose of this study is thus to compare the efficacy of a single pre-operative dose vs a short-term (24-hour) course of cefazolin in preventing SSIs following orthognathic surgery. To our knowledge, no such study has been completed to date. In particular, due to the fact that the vast majority of SSIs following orthognathic surgery occur in the mandible, the investigators will be considering orthognathic surgical procedures including bilateral sagittal split osteotomies, with and without concurrent osteotomies.

Our department's current standardized protocol at the QEII Health Sciences Center for perioperative antibiotic administration is a single pre-operative dose of 2g of cefazolin IV, followed by further doses every 8 hours for a total of 24 hours (3 doses). Here the investigators propose a plan for a prospective, randomized controlled trial comparing this standard regimen to one utilizing a single pre-operative dose of 2g IV cefazolin.

Purpose

To determine the effectiveness of single pre-operative dose vs 24-hour peri-operative IV ampicillin and IV cefazolin in preventing surgical site infection following orthognathic surgery, in particular following bilateral sagittal split osteotomy. The primary outcome of this study is the rate of development of surgical site infection following the described antibiotic protocols. Secondary outcomes are incidence of medication adverse effects, SSI rates in relation to age, sex, smoking status, type of surgery, length of surgery, surgical complications, and medication adverse effects.

Study Design

The aim of this study to conduct a prospective, randomized controlled trial evaluating patients undergoing orthognathic surgery including bilateral sagittal split osteotomies with or without concomitant maxillary and/or chin surgery, with or without wisdom teeth extraction.

The investigators plan to enrol roughly 400 participants in this study. Current literature on antibiotic prophylaxis for orthognathic surgery utilized sample sizes ranging between 30 - 171 participants, with individual group sizes ranging from 14 - 86 participants. Sample size calculation was done based on a study in 2010, comparing single pre-operative dose vs 24-hour peri-operative IV ampicillin. Using a significance level of 5% and a power of 80%, the required sample size was found to be 396 participants when comparing two groups, or 198 participants per group. As such, the investigators will aim to enrol 400 participants. The QEII department of Oral and Maxillofacial Surgery completes roughly 300 orthognathic surgeries per year. The investigators thus anticipate recruitment will continue for 2-3 years. Once data for 30 participants in each group has been gathered, the investigators will analyze this data as a pilot study to re-calculate the sample size needed.

Methodology

All patients meeting the inclusion criteria will be offered participation, and informed consent will be obtained at the pre-operative appointment following surgical consent. The patients will then be assigned a study number and randomly allocated to one of two groups as follows:

A) Single pre-operative dose of 2g IV Cefazolin B) Single pre-operative dose of 2g IV Cefazolin followed by a 24-hour course of 2g IV Cefazolin every 8 hours

Informed consent will be obtained at each participant's pre-operative assessment in the days leading up to the procedure. The discussion will be carried out by the resident conducting the pre-operative assessment, who will have previously completed a training session clarifying the protocol and all aspects of the consent form. Following the informed consent discussion, each new participant will be assigned a study number and asked to select an envelope from a jar which has been sufficiently mixed. Group A or B will be assigned to each study number. Group designations will correspond to a specific protocol, as listed above. The participant's group designation will be documented on the pre-operative assessment sheet. At the time of surgery, the resident completing the post-operative orders will order the corresponding protocol. All orthognathic surgical procedures will then be completed using the standard protocol.

All patients will receive the same post-operative instructions and will be discharged with 0.12% chlorhexidine mouth rinse to be used for 2 weeks following discharge. Patients will return for follow-up at 2 weeks, 4 weeks, and 6 weeks following discharge. Surgical site infection diagnosis will be made according to the CDC criteria and will be reported as either superficial, deep, or organ/space infections. Date of occurrence, location of infection, and treatment provided will be recorded on a standard form provided to each surgeon. Surgeons will be trained prior to commencement of the study regarding CDC criteria and reporting.

For each patient, the osteotomies completed will be documented, along with age, gender, smoking status, length of procedure, and complications. Complications including medication adverse reaction (allergy, toxicity, side effects), surgical complications, and any other significant complications related to the medications or deemed to be relevant to infection risk will be documented. Patients experiencing significant adverse reactions will be instructed to immediately discontinue the causative agent. Data from such cases will be utilized to analyze the rates of adverse effects within each antibiotic regimen. All members of the research team will have access to documentation regarding adverse reactions and will be notified of such events. Significant rates of adverse effects, or serious reactions will prompt a meeting to investigate and discuss further action. Semi-annual reports on adverse events will be prepared and discussed with the research team. The principal investigator will continuously monitor emerging data regarding the efficacy and safety of the agents used in the study. Should any significant issues arise, including unexpected events, serious adverse events, emergent data negatively affecting the safety of the study, privacy breaches, or significant changes to the protocol, this will be reported to the REB. In addition, any data present regarding similar events will be reviewed, and changes to avoid similar situations will be proposed. Should an ongoing concern arise, other participants will be notified, and consent forms will be modified.

At the end of the 6-week data collection period, participant data will be de-identified, and will be designated only by study number. Data from each appointment will initially be in paper format on standard forms. At the end of the 6-week data collection period, data will be converted into electronic format on an excel spreadsheet in de-identified form. The electronic data will be stored via an NSHA computer on the CDHA OMS drive. Paper data will be stored in a filing cabinet in a locked office.

Following data analysis, once data is ready for destruction, 15 years following the completion of the study, the Director of Health Information Services will be contacted, and data will be destroyed as per Nova Scotia Health procedures in a manner that does not allow information to be recognizable, retrievable, readable, or reconstructed. Physical data will be shredded, and electronic data will be deleted with further emptying of "recycle" to facilitate permanent deletion.

Throughout the study, participants will be able to withdraw from the study at any time. Patients will be given a phone number through which they can contact the principal investigator, who will then facilitate the withdrawal. There will be no caveats for withdrawing from the study, and patients will be followed-up as normal.

Data Collection and Analysis

Data will be gathered from patient health questionnaire, inpatient records (anesthesia and nursing records, progress notes, and operative reports), as well as the SSI evaluation form completed at each follow-up appointment. Data collected will include patient age (years), sex, smoking status, osteotomies completed (BSSO with or without other maxillary or mandibular osteotomies), length of procedure in minutes, surgical complications, and medication adverse effects.

The primary outcome will be the rate of surgical site infection utilizing each antibiotic regimen. The secondary outcomes are the incidence of medication adverse effects, and the effect of age, sex, smoking status, completed osteotomies, procedure length, surgical complications, and medication adverse effects on SSI rates.

Data analysis, using longitudinal statistical analysis and inference, to be completed by AI Statistical Solutions, a consulting company operated by professional statisticians Dr. Hong Gu and Dr. Toby Kenney. The investigators plan to utilize generalized linear mixed effect models to test the significance of the infection rates, as well as conclude if there is any relation to age, sex, smoking status, type of surgery, length of surgery, surgical complications, or medication adverse effects. Rates of medication adverse effects will be compared using a z-test or chi-squared test.

Research Ethics

This study will comply with all measures required by the NSHA Research Ethics Board. All protocols have been developed in alignment with guidelines placed by the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use, the Tri-Council Policy Statement: Ethical Conduct for Research Involving Humans (TCPS 2), as well as Division 5 of Health Canada's Food and Drug Regulations.

Confidentiality

Patient information will be secured either on a password protected folder on the hospital network or in a locked office filing cabinet within the department of Oral and Maxillofacial Surgery at the QEII Health Sciences Center. Access will only be given to those directly involved in the study. Data will be de-identified, and each participant will be identified only by a study number. Only necessary data will be stored. Following completion of the study, data will be stored for 15 years, after which the Director of Health Information Services will be contacted, and data will be destroyed as per Nova Scotia Health procedures in a manner that does not allow information to be recognizable, retrievable, readable, or reconstructed.

Informed Consent

Informed consent will be obtained at each participant's pre-operative assessment in the days leading up to the procedure. The discussion will be carried out by the resident conducting the pre-operative assessment, who will have previously completed a training session clarifying the protocol and all aspects of the consent form. The training session will include a discussion of the study design, detailed protocol, as well as a thorough discussion of the consent form. A developed SOP will be provided to each staff member outlining the procedure for obtaining consent, which will also be discussed at the training session. Staff will be given opportunities to ask questions for clarification, and will be given PI contact information should any questions arise. Documentation of training will be completed.

The consent discussion will be carried out in accordance with ICH-GCP guidelines. Investigators and staff conducting the consent discussion will not coerce or influence a patient to participate. Potential participants will be fully informed of all pertinent aspects of the study, and will be provided with a copy of the consent form. Time for inquiry and decision making will be provided to all patients. The discussion will be conducted using simplified language, and all questions will be appropriately answered. The staff member carrying out the discussion will clearly outline the purpose, probability of assignment, subject responsibility, duration of participation, risks, benefits, and that study participation is voluntary, with the choice of withdrawal available at any time. Following the discussion and answering of any questions, the consent form will be signed personally by the participant. The consent form will be updated should any new information available affect patient care or willingness to participate. Any new information that will affect participants already in the study will be communicated to such participants.

Participants will be able to withdraw from the study at any time. Patients will be given a phone number through which they can contact the principal investigator, who will then facilitate withdrawal. There will be no caveats for withdrawing from the study, and patients will be followed-up as normal.

Patient benefits

The potential benefits to participants are dependent largely on the study outcomes. Should one regimen be found to be superior, benefits would include lower rates of complication, morbidity, and healthcare burden. If a lower dose is equally effective, potential benefits would include decreased probability of antibiotic side effects, and decreased development of antibiotic resistance. Potential benefit to future patients undergoing orthognathic surgery if one regimen is found to be superior to the other in preventing surgical site infection.

Patient harms

No significant harms to study participants. Potential harms include allergic reactions to the agents administered, drug toxicity, and secondary infection due to antibiotic use. Standard treatment and monitoring will be employed in the event of allergic reaction. The offending agent will be discontinued immediately if drug toxicity is suspected. Participants may withdraw at any time. Secondary infection will be treated with appropriate antimicrobial administration. Potential increased rate of infection if one regimen is found to be inferior compared to another.

ELIGIBILITY:
Inclusion Criteria:

* All patients ASA 1 and 2 over the age of 16 undergoing orthognathic surgery will be offered participation in this study

Exclusion Criteria:

* Patients ASA 3 and higher, use of antibiotics in the preceding 2 weeks, presence of systemic, oral, or odontogenic infections, patients in a state of immunosuppression as a result of medications or systemic disease, patients with allergies to penicillins or cephalosporins, and patients who lack capacity for informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection Rate | 6 weeks
  Patients will be evaluated at 2, 4, and 6 weeks post-surgery. Surgical sites will be evaluated for presence of infection. Infections will be classified as superficial, deep, or space infection. This information, along with the location of the infection, will be recorded on a standardized form provided to surgeons. Presence of infection will be reported as "yes" or "no". Type of infection will be reported as "superficial", "deep" or "space". Location will be reported as "right maxilla", "left maxilla", "right mandible", or "left mandible".

SECONDARY OUTCOMES:
Rate of Medication Adverse Effects | 6 weeks
  Any observed adverse effect will be documented. For example, if a rash is observed, "rash" will be entered into the "adverse effect" column next to the patient's study number on the data collection sheet. Numbers of "rash" reports will be added to determine the rate of this adverse effect. The total number of all adverse effects will also be added to determine the rate of all adverse effects (%).
Impact of sex on surgical site infection rate | 6 weeks
  The rate of infection (%) in biological male participants will be compared to that in biological female participants to determine if there is any significant difference.
Impact of smoking status on surgical site infection rate | 6 weeks
  The rate of infection (%) in non-smoker participants will be compared to that in smoker participants to determine if there is any significant difference.
Impact of surgery type on surgical site infection rate | 6 weeks
  The rate of infection (%) in participants who had a BSSO alone will be compared to that in participants who had a BSSO in combination with Lefort 1 osteotomies and/or functional genioplasty to determine if there is any significant difference.
Impact of surgical complications on surgical site infection rate | 6 weeks
  The rate of infection (%) in participants who had no surgical complications will be compared to that in participants who had surgical complications to determine if there is any significant difference.
Impact of medication adverse effects on surgical site infection rate | 6 weeks
  The rate of infection (%) in participants who had a medication adverse effect will be compared to that in participants who had no medication adverse effect to determine if there is any significant difference.
Impact of surgery length on surgical site infection rate | 6 weeks
  A linear regression model will be utilized to assess if there is any correlation between length of surgery (minutes) and surgical site infection rate (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria General Hospital, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be useful to be shared.

REFERENCES:
- [Background] Panula K, Finne K, Oikarinen K. Incidence of complications and problems related to orthognathic surgery: a review of 655 patients. J Oral Maxillofac Surg. 2001 Oct;59(10):1128-36; discussion 1137. doi: 10.1053/joms.2001.26704. PMID 11573165
- [Background] Davis CM, Gregoire CE, Steeves TW, Demsey A. Prevalence of Surgical Site Infections Following Orthognathic Surgery: A Retrospective Cohort Analysis. J Oral Maxillofac Surg. 2016 Jun;74(6):1199-206. doi: 10.1016/j.joms.2016.01.040. Epub 2016 Jan 30. PMID 26917207
- [Background] Zijderveld SA, Smeele LE, Kostense PJ, Tuinzing DB. Preoperative antibiotic prophylaxis in orthognathic surgery: a randomized, double-blind, and placebo-controlled clinical study. J Oral Maxillofac Surg. 1999 Dec;57(12):1403-6; discussion 1406-7. doi: 10.1016/s0278-2391(99)90718-8. PMID 10596659
- [Background] Gil APS, Haas OL Jr, Machado-Fernandez A, Munoz-Pereira ME, Velasques BD, da Rosa BM, Favoreto AXP, de Oliveira RB. Antibiotic prophylaxis in orthognathic surgery: an overview of systematic reviews. Br J Oral Maxillofac Surg. 2021 Dec;59(10):1174-1185. doi: 10.1016/j.bjoms.2021.05.010. Epub 2021 May 18. PMID 34465488
- [Background] Danda AK, Ravi P. Effectiveness of postoperative antibiotics in orthognathic surgery: a meta-analysis. J Oral Maxillofac Surg. 2011 Oct;69(10):2650-6. doi: 10.1016/j.joms.2011.02.060. Epub 2011 May 6. PMID 21549486
- [Background] Davis CM, Gregoire CE, Davis I, Steeves TW. Prevalence of Surgical Site Infections Following Orthognathic Surgery: A Double-Blind, Randomized Controlled Trial on a 3-Day Versus 1-Day Postoperative Antibiotic Regimen. J Oral Maxillofac Surg. 2017 Apr;75(4):796-804. doi: 10.1016/j.joms.2016.09.038. Epub 2016 Oct 3. PMID 27789268
- [Background] 7. Jamali, S., Rezaei, F., Pourarz, S., Mohammadi, S. S. M., & Ahmadizadeh, H. (2019). The effect of antibiotics and corticosteroids on orthognathic surgery: a meta-analysis and systematic review. Annals of Medical and Health Sciences Research, 9(1).
- [Background] Tan SK, Lo J, Zwahlen RA. Perioperative antibiotic prophylaxis in orthognathic surgery: a systematic review and meta-analysis of clinical trials. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011 Jul;112(1):19-27. doi: 10.1016/j.tripleo.2010.07.015. Epub 2010 Dec 17. PMID 21168350
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol. 1999 Apr;20(4):250-78; quiz 279-80. doi: 10.1086/501620. No abstract available. PMID 10219875
- [Background] Baqain ZH, Hyde N, Patrikidou A, Harris M. Antibiotic prophylaxis for orthognathic surgery: a prospective, randomised clinical trial. Br J Oral Maxillofac Surg. 2004 Dec;42(6):506-10. doi: 10.1016/j.bjoms.2004.06.010. PMID 15544879
- [Background] Fridrich KL, Partnoy BE, Zeitler DL. Prospective analysis of antibiotic prophylaxis for orthognathic surgery. Int J Adult Orthodon Orthognath Surg. 1994;9(2):129-31. PMID 7989814
- [Background] Jansisyanont P, Sessirisombat S, Sastravaha P, Bamroong P. Antibiotic prophylaxis for orthognathic surgery: a prospective, comparative, randomized study between amoxicillin-clavulanic acid and penicillin. J Med Assoc Thai. 2008 Nov;91(11):1726-31. PMID 19127796
- [Background] Kang SH, Yoo JH, Yi CK. The efficacy of postoperative prophylactic antibiotics in orthognathic surgery: a prospective study in Le Fort I osteotomy and bilateral intraoral vertical ramus osteotomy. Yonsei Med J. 2009 Feb 28;50(1):55-9. doi: 10.3349/ymj.2009.50.1.55. Epub 2009 Feb 24. PMID 19259349
- [Background] Ghantous Y, Araidy S, Yaffe V, Mirochnik R, El-Raziq MA, El-Naaj IA. The efficiency of extended postoperative antibiotic prophylaxis in orthognathic surgery: A prospective, randomized, double-blind, placebo-controlled clinical trial. J Craniomaxillofac Surg. 2019 Feb;47(2):228-232. doi: 10.1016/j.jcms.2018.11.017. Epub 2018 Nov 28. PMID 30578013
- [Background] Tan SK, Lo J, Zwahlen RA. Are postoperative intravenous antibiotics necessary after bimaxillary orthognathic surgery? A prospective, randomized, double-blind, placebo-controlled clinical trial. Int J Oral Maxillofac Surg. 2011 Dec;40(12):1363-8. doi: 10.1016/j.ijom.2011.07.903. Epub 2011 Aug 25. PMID 21871782
- [Background] Eshghpour M, Khajavi A, Bagheri M, Banihashemi E. Value of prophylactic postoperative antibiotic therapy after bimaxillary orthognathic surgery: a clinical trial. Iran J Otorhinolaryngol. 2014 Oct;26(77):207-10. PMID 25320697
- [Background] Danda AK, Wahab A, Narayanan V, Siddareddi A. Single-dose versus single-day antibiotic prophylaxis for orthognathic surgery: a prospective, randomized, double-blind clinical study. J Oral Maxillofac Surg. 2010 Feb;68(2):344-6. doi: 10.1016/j.joms.2009.09.081. PMID 20116706
- [Background] Wahab PU, Narayanan V, Nathan S, Madhulaxmi. Antibiotic prophylaxis for bilateral sagittal split osteotomies: a randomized, double-blind clinical study. Int J Oral Maxillofac Surg. 2013 Mar;42(3):352-5. doi: 10.1016/j.ijom.2012.10.036. Epub 2012 Dec 21. PMID 23265757
- [Background] Ruggles JE, Hann JR. Antibiotic prophylaxis in intraoral orthognathic surgery. J Oral Maxillofac Surg. 1984 Dec;42(12):797-801. doi: 10.1016/0278-2391(84)90348-3. PMID 6594473
- [Background] Bentley KC, Head TW, Aiello GA. Antibiotic prophylaxis in orthognathic surgery: a 1-day versus 5-day regimen. J Oral Maxillofac Surg. 1999 Mar;57(3):226-30; discussion 230-2. doi: 10.1016/s0278-2391(99)90664-x. PMID 10077192
- [Background] Lazzarini L, Brunello M, Padula E, de Lalla F. Prophylaxis with cefazolin plus clindamycin in clean-contaminated maxillofacial surgery. J Oral Maxillofac Surg. 2004 May;62(5):567-70. doi: 10.1016/j.joms.2003.12.004. PMID 15122561
- [Background] Lindeboom JA, Baas EM, Kroon FH. Prophylactic single-dose administration of 600 mg clindamycin versus 4-time administration of 600 mg clindamycin in orthognathic surgery: A prospective randomized study in bilateral mandibular sagittal ramus osteotomies. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2003 Feb;95(2):145-9. doi: 10.1067/moe.2003.54. PMID 12582352
- [Background] Remschmidt B, Schwaiger M, Gaessler J, Wallner J, Zemann W, Schwaiger M. Surgical site infections in orthognathic surgery: prolonged versus single-dose antibiotic prophylaxis. Int J Oral Maxillofac Surg. 2023 Feb;52(2):219-226. doi: 10.1016/j.ijom.2022.06.002. Epub 2022 Jun 25. PMID 35760661
- [Background] Rose J, Crosbie M, Stewart A. A qualitative literature review exploring the drivers influencing antibiotic over-prescribing by GPs in primary care and recommendations to reduce unnecessary prescribing. Perspect Public Health. 2021 Jan;141(1):19-27. doi: 10.1177/1757913919879183. Epub 2019 Oct 21. PMID 31633458
- [Background] Kuriyama T, Karasawa T, Nakagawa K, Saiki Y, Yamamoto E, Nakamura S. Bacteriologic features and antimicrobial susceptibility in isolates from orofacial odontogenic infections. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2000 Nov;90(5):600-8. doi: 10.1067/moe.2000.109639. PMID 11077383
- [Background] Poeschl PW, Spusta L, Russmueller G, Seemann R, Hirschl A, Poeschl E, Klug C, Ewers R. Antibiotic susceptibility and resistance of the odontogenic microbiological spectrum and its clinical impact on severe deep space head and neck infections. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Aug;110(2):151-6. doi: 10.1016/j.tripleo.2009.12.039. Epub 2010 Mar 25. PMID 20346713
- [Background] Kuriyama T, Karasawa T, Nakagawa K, Yamamoto E, Nakamura S. Incidence of beta-lactamase production and antimicrobial susceptibility of anaerobic gram-negative rods isolated from pus specimens of orofacial odontogenic infections. Oral Microbiol Immunol. 2001 Feb;16(1):10-5. doi: 10.1034/j.1399-302x.2001.160102.x. PMID 11169133
- [Background] Harrison CJ, Bratcher D. Cephalosporins: a review. Pediatr Rev. 2008 Aug;29(8):264-7; quiz 273. doi: 10.1542/pir.29-8-264. No abstract available. PMID 18676578
- [Background] Brook I, Wexler HM, Goldstein EJ. Antianaerobic antimicrobials: spectrum and susceptibility testing. Clin Microbiol Rev. 2013 Jul;26(3):526-46. doi: 10.1128/CMR.00086-12. PMID 23824372
- [Background] Heim N, Faron A, Wiedemeyer V, Reich R, Martini M. Microbiology and antibiotic sensitivity of head and neck space infections of odontogenic origin. Differences in inpatient and outpatient management. J Craniomaxillofac Surg. 2017 Oct;45(10):1731-1735. doi: 10.1016/j.jcms.2017.07.013. Epub 2017 Jul 28. PMID 28838838
- [Background] 32. Abdulla, A. H. Identification and Antimicrobial Susceptibility of Bacterial Isolates from Odontogenic Abscesses.